CLINICAL TRIAL: NCT02117713
Title: A Multicenter Extension Study to Evaluate the Long-Term Safety and Durability of the Therapeutic Effect of LUM001, an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi), in the Treatment of Cholestatic Liver Disease in Pediatric Subjects With Alagille Syndrome
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Durability of Effect of LUM001 in the Treatment of Cholestatic Liver Disease in Pediatric Subjects With Alagille Syndrome
Acronym: IMAGINE-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Collaborators: Lumena Pharmaceuticals, Inc. (Industry); Childhood Liver Disease Research and Education Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LUM001-305; SHP625-305 (Other: Shire)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome | interventions — maralixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM001 (Maralixibat) (Experimental): Participant will receive LUM001 also known as Maralixibat (MRX) administered orally once per day.
  Interventions: Drug: LUM001 (Maralixibat)

INTERVENTIONS:
Drug: LUM001 (Maralixibat) — Dosing of LUM001 also known as Maralixibat (MRX) with the objective of achieving optimal control of pruritus at a dose level that is tolerated by the participant and up to a maximum daily dose of 280 micrograms per kilogram (mcg/kg).

SUMMARY:
This is a multicentre, extension study of LUM001 in children diagnosed with Alagille Syndrome who have completed participation in a core LUM001 treatment protocol. The primary objective is to evaluate long-term safety and tolerability of LUM001. Efficacy will be assessed by evaluating the effect of LUM001 on the biochemical markers and pruritus associated with Alagille Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 12 months to 18 years of age.
2. Competent to provide informed consent and assent (per institutional review board/Ethics Committee [IRB/EC]), as appropriate.
3. Completed participation in the LUM001-301 protocol.
4. Females of childbearing potential must have a negative urine pregnancy test [beta human chorionic gonadotropin (beta-hCG)] at the Baseline Visit.
5. Sexually active females must be prepared to use an effective method of contraception during the trial.

   Effective methods of contraception are considered to be:
   1. Hormonal (for example, contraceptive pill, patch, intramuscular implant or injection); or
   2. Barrier method, for example, (a) condom with spermicide, or (b) diaphragm, with spermicide; or
   3. Intrauterine device (IUD).
6. Participants above the age of assent and caregivers and children must be able to read and understand English or Spanish.
7. Caregivers (and age appropriate participants) must have access to phone for scheduled calls from study site.
8. Caregivers (and age appropriate participants) must be willing and able to complete a daily electronic diary (ItchRO) during the first consecutive 12 weeks of the study and then for 4 consecutive weeks following the Week 24 and Week 44 visits.
9. Caregivers (and age appropriate participants) must digitally accept the licensing agreement in the ItchRO electronic diary software at the outset of the study.
10. Eligible participants must be able to adhere to local Ethics Committee or Institutional Review Board (IRB) blood volume limits for laboratory testing.
11. The participant has completed the protocol either through Week 144, or the End of Trial visit, or has received permission from the sponsor and the Premier Medical monitor to re-enter the study in the long-term, optional follow-up treatment period 2.
12. Females of child-bearing potential must have a negative urine or serum pregnancy test (beta-HCG]) at the time of entry into the long-term optional follow-up treatment period 2.
13. Male and female participants of child-bearing potential who are sexually active, or are not currently sexually active, but become sexually active during the study or for 30 days following the last dose of study drug, must agree to use acceptable contraception during the study.
14. Informed consent and assent (per IRB/EC) as appropriate.
15. Caregivers (and age appropriate participants) must have access to phone for scheduled calls from study site.
16. Caregivers (and age appropriate participants) must be willing to follow the rules of eDiary completion.

Exclusion Criteria:

1. Experienced an adverse event or serious adverse event (SAE) related to the study drug during the LUM001-301 protocol that led to the discontinuation of the participant from the core study.
2. Any conditions or abnormalities (including laboratory abnormalities) which in the opinion of the Investigator, Medical Monitor or ChiLDReN Protocol Chair, may compromise the safety of the participant, or interfere with the participant participating in or completing the study.
3. History or known presence of gallstones or kidney stones.
4. History of non-adherence during the participant's participation in the LUM001-301 protocol. Non-adherence is defined by dosing compliance (dosing compliance is calculated by [the total number of doses that were actually taken by the participant] divided by [the total number of doses that should have been taken by the participant] multiplied by 100) of less than 80% in the LUM001-301 protocol.
5. Unlikely to comply with the study protocol, or unsuitable for any other reason, as judged by the investigator.
6. All above exclusion criteria will apply upon re-entry into the long-term, optional follow-up treatment period 2.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (11):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at San Francisco Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LUM001 (Maralixibat): Participant received LUM001 also known as Maralixibat (MRX) administered orally once per day for up to 216 weeks.
Period: Week 48
Arm/Group | LUM001 (Maralixibat)
Started | 34
Completed | 26
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Withdrawal by caregiver | 2
Not completed — Did not consent to Protocol Amendment 4 | 2
Period: Long Term Follow-up Treatment
Arm/Group | LUM001 (Maralixibat)
Started | 26
Completed | 20
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Progressive Disease | 2
Not completed — Non-Compliance with study drug | 1

BASELINE CHARACTERISTICS:
Population: In the lead-in Study LUM001-301, participants were randomized to receive either placebo or active drug (MRX). The last observation obtained before first dose of MRX (either for participants who received MRX or placebo LUM001-301) was used as the MRX baseline observation for all calculations of change. For participants who were assigned MRX in LUM001-301, results at each post-baseline analysis visit included up to 13 more weeks of treatment than participants who were assigned placebo.
Groups:
- Core Study Period: Participant received LUM001 also known as Maralixibat (MRX) administered orally once per day.
Arm/Group | Core Study Period
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years of age] | 7 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From MRX Baseline to Week 48 in Fasting Serum Bile Acid (sBA)
Description: This primacy efficacy endpoint is the mean change from MRX baseline to week 48 in fasting sBA levels.
Time Frame: Baseline to Week 48
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- MRX Baseline Value: These are the MRX baseline values for participants
- Maralixibat Week 48 Values: Week 48 values for participants.
Arm/Group | MRX Baseline Value | Maralixibat Week 48 Values
Number analyzed (Participants) | 34 | 26
μmol/L | 223.62 (205.041) | 157.35 (178.538)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Maralixibat Week 48 Values; Test type: Equivalence — Student's t-test used to test if mean change is statistically significant; null hypothesis is that the mean change from baseline is equal to zero; p = 0.1157, Student's t-test; Mean Difference (Net) = -28.59, 95% CI 2-sided [-64.72 to 7.54], Standard Deviation 89.456 — Difference is only calculated in participants who had baseline and week 48 values for n= 26

2. Secondary Outcome: Change From MRX Baseline to Week 216 in Fasting Serum Bile Acid (sBA)
Description: The secondary endpoint of this study was the mean change from MRX baseline to week 216 fasting in sBA levels.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Maralixibat Baseline Values: These are the MRX baseline values for participants.
- Week 216: These are the week 216 values of participants
Arm/Group | Maralixibat Baseline Values | Week 216
Number analyzed (Participants) | 34 | 10
μmol/L | 223.62 (205.041) | 118.81 (126.878)
Statistical Analysis 1: Comparison: Maralixibat Baseline Values vs Week 216; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1469, Student's t-test; Mean Difference (Net) = -45.15, 95% CI 2-sided [-109.48 to 19.19], Standard Deviation 89.934; Difference is only calculated in participants who had baseline and week 216 values for n=10

3. Secondary Outcome: Change From Baseline to Week 218 in Pruritus
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time to week 218 in pruritus as measured by ItchRO(Obs) weekly average morning severity score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe). Results reported here are the long-term results.
Time Frame: Baseline to Week 218
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Week 218: These are values from Week 218.
Arm/Group | Maralixibat Baseline Values | Week 218
Number analyzed (Participants) | 34 | 6
score on a scale | 2.533 (0.8423) | 0.429 (0.8571)
Statistical Analysis 1: Comparison: Maralixibat Baseline Values vs Week 218; Test type: Equivalence — Student's t-test was used to test if mean change was statistically significant (null hypothesis is that the mean change from baseline is equal to zero); p = 0.005, Student's t-test; Mean Difference (Net) = -2.353, 95% CI 2-sided [-3.101 to -1.606], Standard Deviation 0.7124 — Difference is only calculated in participants who had baseline and week 218 values for n=6

4. Secondary Outcome: Change From Baseline to Week 216 in Alanine Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in ALT levels.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Week 216 Values: These are the week 216 values for participants.
Arm/Group | MRX Baseline Value | Week 216 Values
Number analyzed (Participants) | 34 | 7
U/L | 152.9 (82.26) | 222.4 (126.53)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216 Values; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.2607, Student's t-test; Mean Difference (Net) = 56.0, 95% CI 2-sided [-54.4 to 166.4], Standard Deviation 119.32 — Difference is only calculated in participants who had baseline and week 216 values for n=7

5. Secondary Outcome: Change From Baseline to End of Treatment in Alkaline Phosphatase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in ALP levels.
Time Frame: Baseline to Week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Week 216 Values: These are the 2616 values for participants.
Arm/Group | MRX Baseline Value | Week 216 Values
Number analyzed (Participants) | 34 | 7
U/L | 598.8 (199.89) | 528.3 (221.93)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216 Values; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.1340, Student's t-test; Mean Difference (Net) = -141.6, 95% CI 2-sided [-341.6 to 58.4], Standard Deviation 216.25 — Difference is only calculated in participants who had baseline and week 216 values for n=7

6. Secondary Outcome: Change From MRX Baseline to Week 216 in Aspartate Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in AST levels.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Week 216: These are the week 216 values for participants.
Arm/Group | MRX Baseline Value | Week 216
Number analyzed (Participants) | 34 | 7
U/L | 149.7 (88.27) | 231.4 (122.26)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.1474, Student's t-test; Mean Difference (Net) = 47.6, 95% CI 2-sided [-22.4 to 117.6], Standard Deviation 75.68 — Difference is only calculated in participants who had baseline and week 216 values for n=7

7. Secondary Outcome: Change From MRX Baseline to Week 216 in Clinician Xanthoma Severity Score
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in clinician xanthoma severity scores. It is based on a 0-4 scale to rate the number of lesions present and the degree to which the lesions interfere or limit activities. Clinician xanthoma severity scores range from 0 to 4, with a score of zero representing no evidence of xanthomatosis and a score of 4 representing xanthoma so severe that it is disabling.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | MRX Baseline Value | Week 216
Number analyzed (Participants) | 34 | 7
Points | 0.9 (1.33) | 1.1 (1.68)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 1.00, Student's t-test; Mean Difference (Net) = 0, 95% CI 2-sided [-0.5 to 0.5], Standard Deviation 0.58 — Difference is only calculated in participants who had baseline and week 216 values for n=7

8. Secondary Outcome: Change From Baseline to Week 216/LOFC Clinician Scratch Scale (CSS) Score
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time to week 216/LOCF in pruritus as measured by the Clinician Scratch Scale (CSS). The Clinician Scratch Scale uses a 5-point scale, where 0 = none; 1 = rubbing or mild scratching when undistracted; 2 = active scratching without evident skin abrasions; 3 = abrasion evident; 4 = cutaneous mutilation, haemorrhage and scarring evident.
Time Frame: Baseline to Week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | MRX Baseline Value | Week 216
Number analyzed (Participants) | 34 | 7
Points | 2.9 (1.08) | 1.1 (1.07)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216; Test type: Equivalence — Student's t-test used to test if mean change is statistically significant (null hypothesis is that the mean change from baseline is equal to zero); p = 0.0167, Student's t-test; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3 to -0.4], Standard Deviation 1.38 — Difference is only calculated in participants who had baseline and week 216 values for n=7

9. Secondary Outcome: Change From MRX Baseline to Week 216 in Gamma Glutamyltransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in GGT.
Time Frame: Baseline to Week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Week 216 Values: These are the week 216 values of the participants.
Arm/Group | MRX Baseline Value | Week 216 Values
Number analyzed (Participants) | 34 | 7
U/L | 493.5 (380.29) | 431 (235.35)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216 Values; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.9108, Student's t-test; Mean Difference (Net) = 10.9, 95% CI 2-sided [-216.6 to 238.3], Standard Deviation 245.92 — Difference is only calculated in participants who had baseline and week 216 values for n=7

10. Secondary Outcome: Mean Change From MRX Baseline to Week 216 in Total Bilirubin
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in total bilirubin.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MRX Baseline Value | Week 216
Number analyzed (Participants) | 34 | 7
mg/dL | 5.62 (6.420) | 5.39 (5.181)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216; Test type: Equivalence — Student's t-test was used to test if mean change was statistically significant(null hypothesis is that the mean change from baseline is equal to zero); p = 0.1207, Student's t-test; Mean Difference (Net) = 0.1207, 95% CI 2-sided [-3.03 to 0.45], Standard Deviation 1.882 — Difference is only calculated in participants who had baseline and week 216 values for n=7

11. Secondary Outcome: Mean Change From MRX Baseline to Week 216 in Direct Bilirubin
Description: This secondary efficacy endpoint is the mean change from MRX baseline to week 216 in direct bilirubin.
Time Frame: Baseline to week 216
Population: Since most participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MRX Baseline Value | Week 216 Values
Number analyzed (Participants) | 34 | 7
mg/dL | 3.541 (3.6433) | 3.714 (3.8369)
Statistical Analysis 1: Comparison: MRX Baseline Value vs Week 216 Values; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0927, Student's t-test; Mean Difference (Net) = -0.943, 95% CI 2-sided [-2.098 to 0.212], Standard Deviation 1.2488 — Difference is only calculated in participants who had baseline and week 216 values for n=7

ADVERSE EVENTS:
Time Frame: Baseline to End of Treatment (Week 216)
Groups:
- LUM001 (Maralixibat): Participant received LUM001 (also known as Maralixibat or MRX) as oral solution once daily based on participant's weight. The dose was escalated from 14, 35, 70, 140 and 280 microgram per kilogram per day (mcg/kg/day) for 4-week dose escalation period. During 8-weeks of dose optimization period, drug was adjusted in titrated manner and dosing was continued to complete the stable dosing and safety monitoring periods for up to 96 weeks of cumulative LUM001 exposure in this study. Dosing during long-term optional follow-up treatment periods 1 and 2 was maintained at the same dose levels as at weeks 96 and 144 for participants rolling over into these treatment periods respectively.
Arm/Group | LUM001 (Maralixibat)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 6/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM001 (Maralixibat) (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM001 (Maralixibat) (N=34)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1 (1)
Non-compaction cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (5)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (2)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (39)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (18)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 13 (37)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Post-tussive vomiting (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (17)
Asthenia (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Fatigue (General disorders) | 1 (1)
Influenza like illness (General disorders) | 6 (22)
Medical device pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 15 (39)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Adenovirus infection (Infections and infestations) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 7 (15)
Ear infection bacterial (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 4 (5)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (2)
Herpes simplex (Infections and infestations) | 1 (5)
Influenza (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (24)
Oral herpes (Infections and infestations) | 1 (2)
Otitis media (Infections and infestations) | 1 (3)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 5 (10)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 6 (11)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (63)
Urinary tract infection (Infections and infestations) | 3 (5)
Viral infection (Infections and infestations) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural anxiety (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (8)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Sports injury (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase abnormal (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (14)
Aspartate aminotransferase abnormal (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Blood albumin increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood bicarbonate decreased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Gamma-glutamyltransferase abnormal (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Heart rate irregular (Investigations) | 1 (1)
International normalised ratio abnormal (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 7 (9)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Ultrasound liver abnormal (Investigations) | 1 (1)
Vitamin D decreased (Investigations) | 2 (3)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (6)
Vitamin E deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin K deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (9)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (16)
Migraine (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Chromaturia (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1)
Adenoidal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (84)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 7 (10)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Xanthoma (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT02117713/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT02117713/SAP_001.pdf